CLINICAL TRIAL: NCT01719133
Title: Détermination de la réactivité cutanée de Volontaires Allergiques au Pollen de Bouleau Contre Des Peptides dérivés de Bet v 1
Brief Title: Skin Prick Tests With AllerT in Subjects Allergic to Birch Pollen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anergis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AN002
Record Dates: First submitted 2012-10-26; First posted 2012-11-01 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Allergic Rhinitis
Keywords: allergy; birch
MeSH Terms: conditions — Rhinitis, Allergic; Hypersensitivity | interventions — Sodium Chloride; Histamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Other): placebo histamine T1 T2 T3 T4 T5 T1-T2-T3 T4-T5
  Interventions: Drug: placebo; Drug: Histamine; Drug: AllerT1; Drug: AllerT2; Drug: AllerT3; Drug: AllerT4; Drug: AllerT5; Drug: mix of AllerT1-T2-T3; Drug: mix of AllerT4-T5

INTERVENTIONS:
Drug: placebo — saline solution
  Other Names: saline
Drug: Histamine — positive control
  Other Names: Histamine solution
Drug: AllerT1 — synthetic peptide T1
Drug: AllerT2 — synthetic peptide T2
Drug: AllerT3 — synthetic peptide T3
Drug: AllerT4 — synthetic peptide T4
Drug: AllerT5 — synthetic peptide T5
Drug: mix of AllerT1-T2-T3 — mix of peptides T1, T2 and T3
  Other Names: AllerT
Drug: mix of AllerT4-T5 — mix T4-T5
  Other Names: mix T4-T5

SUMMARY:
Assessment of skin reactivity by skin prick tests to synthetic peptides derived from the major birch allergen bet v 1, in subjects allergic to birch pollen.

DETAILED DESCRIPTION:
The study tested - all by skin tests - in the same group of 20 trial subjects, one positive control (histamine solution), one negative control (placebo saline) and five experimental peptides called T1, T2, T3, T4 and T5. Results of the skin prick tests were scored as negative (no reaction) or positive (wheal diameter > 4 mm with erythema)

ELIGIBILITY:
Inclusion Criteria:

* history of allergy symptoms during previous birch pollen season
* positive skin prick test to birch pollen extract

Exclusion Criteria:

* pregnancy
* uncontrolled asthma
* other significant clinical conditions or immune disorders
* subjects taking antihistamines or drugs with antihistamine activity

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
skin prick test reactivity | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Francois Spertini, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

REFERENCES:
- [Derived] Pellaton C, Perrin Y, Boudousquie C, Barbier N, Wassenberg J, Corradin G, Thierry AC, Audran R, Reymond C, Spertini F. Novel birch pollen specific immunotherapy formulation based on contiguous overlapping peptides. Clin Transl Allergy. 2013 Jun 1;3(1):17. doi: 10.1186/2045-7022-3-17. PMID 23725004